CLINICAL TRIAL: NCT05784701
Title: Age-descending, Randomized, Placebo-controlled Phase 2 Trial in Three Sites in Sub-Saharan Africa to Assess the Safety and Immunogenicity of a Parenteral Trivalent Salmonella (S. Enteritidis/S. Typhimurium/S. Typhi Vi) Conjugate Vaccine (TSCV) Versus Placebo
Brief Title: Trivalent Salmonella Conjugate Vaccine (TSCV)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Bharat Biotech International (Unknown); Wellcome Trust (Other)
Responsible Party: Principal Investigator, Milagritos Tapia, Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: HP-00103997
Record Dates: First submitted 2023-02-07; First posted 2023-03-27 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Trivalent Salmonella Conjugate Vaccine (TSCV)
Keywords: S. Enteritidis; S. Typhimurium; S. Typhi Vi; Trivalent Salmonella Conjugate Vaccine (TSCV)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- TSCV (Full-strength) (Active Comparator): Full-strength GMP formulation of Trivalent Salmonella Conjugate Vaccine (TSCV)
  Interventions: Drug: TSCV (Full-strength)
- TSCV (Half-strength) (Active Comparator): Half-strength GMP formulation of TSCV
  Interventions: Drug: TSCV (Half-strength)
- Typbar-TCV (Active Comparator): Licensed Monovalent Typbar-TCV
  Interventions: Drug: Typbar-TCV
- Placebo (Placebo Comparator): PBS
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TSCV (Full-strength) — TSCV (Full-strength)
  Arms: TSCV (Full-strength)
Drug: TSCV (Half-strength) — TSCV (Half-strength)
  Arms: TSCV (Half-strength)
Drug: Typbar-TCV — Typbar-TCV
  Arms: Typbar-TCV
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This is an age-descending, randomized, placebo-controlled trial that will evaluate the safety and immunogenicity of a Trivalent Salmonella conjugate vaccine (TSCV). The trial will proceed from adults, to children, to toddlers, and then to infants.

DETAILED DESCRIPTION:
This is an age-descending, randomized, placebo-controlled trial that will evaluate the safety and immunogenicity of a Trivalent Salmonella conjugate vaccine (TSCV). The trial will proceed from adults, to children, to toddlers, and then to infants.

In Step 1A-D of the trial, participants will be randomized to receive a single dose of TSCV (Full-strength or Half-strength), Typbar-TCV, or placebo, first in adults, then in children 5 to 9 years of age, then children 24 to 59 months of age, and then 16 to 23 months of age.

Participants will be followed for 6 months. After a Data Safety Monitoring Board (DSMB) review of the safety data, the trial will proceed to Step 2A and 2B whereupon 12- to 16-month-old toddlers and infants 8- to 11-months of age will be similarly and simultaneously randomized. Participants will be followed for 6 months.

After another DSMB safety review, Step 3 will commence with simultaneous enrollment of 12- to 14-week-old and 16- to 18-week-old infants who will each receive a single dose of TSCV, TCV or placebo. Participants will be followed for 6 months.

After a third DSMB safety review and selection of the preferred TSCV formulation (Full-strength versus Half-strength) for further clinical development (a decision taken by the Sponsor, Manufacturer, and funder, while taking into consideration the recommendation of the DSMB), Step 4 will evaluate a two-dose regimen. Infants 12 to 18 weeks of age will be randomized to receive either two doses of TSCV (at Full-strength or Half-strength, based on results from Steps 1-3) or placebo followed by Typbar-TCV. The priming dose will be administered at enrollment and the booster at ~9, ~12, or ~15-17 months of age.

Participants will be followed until 6 months after the last study vaccination.

Note -- Whenever investigational products are intended to be administered at a scheduled Expanded Program on Immunization visit, they will always be given 2 weeks after the routine EPI vaccines. This will not only avoid interference with EPI vaccines but will provide a convenient contact point for potential recruitment of participants for the study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals, female or male
* Age (all age ranges are inclusive)

  1. Step 1A: Adults 20-35 years of age
  2. Step 1B: Children, 5-9 years of age
  3. Step 1 C: Pre-school children, 24-59 mos. of age
  4. Step 1D: Older toddlers, 16-23 months of age
  5. Step 2A: Young toddlers, 12-16 months of age
  6. Step 2B: Older infants, 8-11 months of age
  7. Step 3: Young infants,12-14 weeks of age OR 16-18 weeks of age
  8. Step 4: Young infants, 12-18 weeks of age
* For potential pediatric participants, the parents must live within the catchment area of the clinical study facility at the time of the study vaccinations and must intend to continue to reside in the area for the duration of the study
* Adult subjects and parents/ guardians of pediatric subjects must have provided informed consent
* Infant and toddler subjects in Steps 2, 3, and 4 must have received their scheduled EPI vaccines at least 14 days prior to receiving a study product.

Exclusion Criteria:

* A history of documented hypersensitivity to any component of the Trivalent Salmonella Conjugate Vaccine or of Typbar-TCV™
* A history of previous vaccination with any licensed or experimental typhoid vaccine A known history of diabetes, tuberculosis, malignancy, chronic kidney disease, cardiac disease, liver disease, progressive neurological disorder, poorly controlled seizure disorder, or a terminal illness based on participant interview and review of screening laboratory results.
* Severe malnutrition: i.e., weight-for-length Z-score of less than - 3.
* Receipt of any other investigational intervention in the last 6 months
* Known HIV infection or other forms of immunocompromise
* Receipt of systemic immunosuppressive medication including systemic corticosteroids
* For Step 1A, for females of child-bearing potential, a positive pregnancy test at the time of enrollment.
* For Step 1B, any female child who has experienced menarche.
* Acute illness with or without fever (temperature >38.0oC) is a temporary exclusion criterion. Enrollment may be postponed until 3 days after the illness has resolved.
* Positive malaria test is a temporary exclusion criterion. Participant may be enrolled 3 days after completing treatment.
* Any condition determined by the investigators to be likely to interfere with evaluation of the vaccine, to be a significant health risk to the participant, or to make it unlikely that the participant would complete the study

Ages: 12 Weeks to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 800 (Estimated)
Dates: Start 2023-04-05 (Actual); Primary Completion 2027-01-05 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Safety and reactogenicity of Full-strength and Half-strength TSCV | first 30 minutes after parenteral immunization
  The proportion of participants in each product group and within each age group who develop adverse events (AEs) in the first 30 minutes after parenteral immunization
Safety and reactogenicity of Full-strength and Half-strength TSCV | over 7 days post-vaccination.
  The proportion of participants in each product group and within each age group who develop adverse events (AEs) in the 7 days post-vaccination.
Safety and reactogenicity of Full-strength and Half-strength TSCV | through Day 29 of follow-up post-vaccination
  The proportion of participants who experience AEs through Day 29 of follow-up post-vaccination.
Safety and reactogenicity of Full-strength and Half-strength TSCV | Through Day 366 of follow-up post vaccination
  The proportion of participants who experience Serious Adverse Events through their participation in the study.
Non-inferiority analysis: immunogenicity of Full-strength vs. Half-strength TSCV | Through day 29 post vaccination
  Serum IgG anti-COPS antibodies (to both S. Enteritidis and S. Typhimurium antigens)
Non-inferiority analysis: immunogenicity of Full-strength vs. Half-strength TSCV | Through day 29 post vaccination
  Serum IgG anti-Vi antibodies
Safety and reactogenicity after primary dose of TSCV and after booster dose of TSCV or Typbar-TCV™ [At each booster age group (9, 12, or 15-17 mo. of age)] | over 7 days post-vaccination.
  The proportion of participants in each product group who develop adverse events (AEs) in 7 days post-vaccination.
Safety and reactogenicity after primary dose of TSCV and after booster dose of TSCV or Typbar-TCV™ [At each booster age group (9, 12, or 15-17 mo. of age)] | through Day 29 of follow-up after each vaccination.
  The proportion of participants who experience AEs through Day 29 of follow-up after each vaccination.
Safety and reactogenicity after primary dose of TSCV and after booster dose of TSCV or Typbar-TCV™ [At each booster age group (9, 12, or 15-17 mo. of age)] | Until the end of the participant study period - 6 months to 1 year post vaccination
  The proportion of participants who experience Serious Adverse Events through their participation in the study.
Immunogenicity of two-dose regimen of TSCV [At each booster age group (9, 12 or 15-17 months of age)] | At day 29 post booster vaccination
  The rates of seroconversion of serum IgG anti-COPS at each booster age group
Immunogenicity of two-dose regimen of TSCV [At each booster age group (9, 12 or 15-17 months of age)] | At day 29 post booster vaccination
  The geometric mean titers of serum IgG anti-COPS at each booster age group
Immunogenicity of two-dose regimen of TSCV [At each booster age group (9, 12 or 15-17 months of age)] | At day 29 post booster vaccination
  The increases in geometric mean-fold titers from day 1 to 29 of serum IgG anti-COPS at each booster age group
Immunogenicity of two-dose regimen of TSCV [At each booster age group (9, 12 or 15-17 months of age)] | At day 29 post booster vaccination
  The rates of persisting seroconversion (titers remaining > 4-fold above Day 1) of serum IgG anti-COPS at each booster age group
Immunogenicity of two-dose regimen of TSCV [At each booster age group (9, 12 or 15-17 months of age)] | At day 29 post booster vaccination
  The rates of seroconversion of serum IgG anti-Vi at each booster age group
Immunogenicity of two-dose regimen of TSCV [At each booster age group (9, 12 or 15-17 months of age)] | At day 29 post booster vaccination
  The geometric mean titers of serum IgG anti-Vi at each booster age group
Immunogenicity of two-dose regimen of TSCV [At each booster age group (9, 12 or 15-17 months of age)] | At day 29 post booster vaccination
  The increases in geometric mean-fold titers from day 1 to 29 of serum IgG anti-Vi at each booster age group
Immunogenicity of two-dose regimen of TSCV [At each booster age group (9, 12 or 15-17 months of age)] | At day 29 post booster vaccination
  The rates of persisting seroconversion (titers remaining > 4-fold above Day 1) of serum IgG anti-Vi at each booster age group

CONTACTS AND LOCATIONS:
Overall Officials: Miligritos Tapia, MD, Principal Investigator — University of Maryland Center for Vaccine Development
Locations (1):
- Centre for Vaccine Development (CVD-Mali), Bamako, Mali

IPD SHARING:
Plan to Share IPD: No